CLINICAL TRIAL: NCT02942641
Title: Indwelling Urinary Catheterization Versus Clean Intermittent Catheterization for the Short-term Management of Hospitalized Patients With Transient Acute Urinary Retention: A Prospective Randomized Trial
Brief Title: Indwelling Urinary Catheterization Versus Clean Intermittent Catheterization for the Short-term Management of Hospitalized Patients With Transient Acute Urinary Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Dr. Pocharapong Jenjitranant, Dr. Pocharapong Jenjitranant, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 095920
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Retention
Keywords: Urethral catheter; clean intermittent catheterization; UTI; pain; quality of life; hematuria; cloudy urine
MeSH Terms: conditions — Urinary Retention; Pain; Hematuria | interventions — Intermittent Urethral Catheterization; Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indwelling urethral catheterization (Foley) (Experimental): Foley catheter as the intervention.
  Interventions: Procedure: Indwelling urethral catheterization (Foley); Device: Foley
- Clean intermittent catheterization (CIC) (Experimental): CIC as the intervention .
  Interventions: Procedure: Clean intermittent catheterization (CIC)

INTERVENTIONS:
Procedure: Indwelling urethral catheterization (Foley) — Hospitalized patients who developed first-time AUR were randomly divided into two groups depending on the type of assigned intervention: CIC and indwelling urethral catheter groups.
  Patients in this group received indwelling urethral catheter as the intervention.
  Arms: Indwelling urethral catheterization (Foley)
Procedure: Clean intermittent catheterization (CIC) — Hospitalized patients who developed first-time AUR were randomly divided into two groups depending on the type of assigned intervention: CIC and indwelling urethral catheter groups.
  Patients in this group received CIC as the intervention.
  Arms: Clean intermittent catheterization (CIC)
Device: Foley
  Arms: Indwelling urethral catheterization (Foley)

SUMMARY:
Objective: Acute urinary retention (AUR) is a common problem in hospitalized patients. Either indwelling urethral catheterization or clean intermittent catheterization (CIC) can be the choice of treatment. In chronic urinary retention, most physicians prefer CIC to chronic indwelling urethral catheter on the basis of the claim that the rate of catheter-associated urinary tract infection (CAUTI) is lower.

Method: The patients were randomized into indwelling urethral catheter and CIC groups. The primary outcomes of the study were catheter-associated asymptomatic bacteriuria and CAUTI. The secondary outcomes were pain, hematuria, cloudy urine, and quality of life.

DETAILED DESCRIPTION:
We queried the hospitalized patients in Ramathibodi Hospital who developed first-time AUR from June 2014 to May 2015. Patients under 18 years of age with a history of urinary retention, urinary tract infection, and poor compliance were excluded from this study. All the patients gave their written informed consents. The patients were randomly divided into two groups depending on the type of assigned intervention: CIC and indwelling urethral catheter groups.

All the patients were followed up after 2 weeks; urinalysis and urine culture were obtained at the time of AUR and whenever the patients developed UTI-associated symptoms. The patients with positive urine culture at the time of AUR were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients in Ramathibodi Hospital who developed first-time AUR from June 2014 to May 2015.

Exclusion Criteria:

* Patients under 18 years of age
* History of urinary retention
* Urinary tract infection
* Poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Catheter-associated urinary tract infection (CAUTI) | up to 12 months
  the presence of symptoms or signs compatible with UTI and no other identified source of infection, along with ≥103 CFU/mL of ≥1 bacterial species in a single catheter urine specimen or in a midstream voided urine specimen from a patient whose urethral catheter has been removed within the previous 48 hours.

SECONDARY OUTCOMES:
Pain | up to 12 months
  Using visual analogue scales
Hematuria | up to 12 months
Cloudy urine | up to 12 months
Quality of life | up to 12 months
  assessed on the basis of social functioning (SF) that was derived from SF-36 questionnaire
Catheter-associated asymptomatic bacteriuria | up to 12 months
  the presence of ≥105 CFU/mL of ≥1 bacterial species in a single catheter urine specimen from a patient without symptoms compatible with UTI.

IPD SHARING:
Plan to Share IPD: Undecided